CLINICAL TRIAL: NCT07148921
Title: Changes in Pain and Perception Thresholds Due to Gender Affirming Hormone Therapy: a Prospective Exploratory Cohort Study
Brief Title: Perception of Pain During Gender Affirming Hormone Therapy
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Oliver Kimberger, Univ. Prof. PD Dr., Medical University of Vienna
Other Study IDs: 1103/2024
Record Dates: First submitted 2025-04-24; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Transgender Persons; Pain Threshold; Perception of Pain; Sex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AFAB Group: Transgender men and transmasculine individuals
  Interventions: Diagnostic Test: Quantitative Sensory Testing; Diagnostic Test: Patient Health Questionnaire 9; Diagnostic Test: Hormone concentrations
- AMAB Group: Transgender women and transfeminine individuals
  Interventions: Diagnostic Test: Quantitative Sensory Testing; Diagnostic Test: Patient Health Questionnaire 9; Diagnostic Test: Hormone concentrations

INTERVENTIONS:
Diagnostic Test: Quantitative Sensory Testing — Quantitative sensory testing (QST) is a psychophysical test procedure. With the help of calibrated stimuli and subjective sensory information, the functional state of the somatosensory system of a subject or patient is examined with regard to the expression of clinical signs.
  The test includes:
  * Cold detection threshold
  * Warm detection threshold
  * Paradoxical heat sensation
  * Cold pain threshold
  * Heat pain threshold
  * Mechanical detection threshold
  * Mechanical pain threshold
  * Mechanical pain sensitivity
  * Dynamic mechanical allodynia
  * Wind-up phenomena
  * Vibration threshold
  * Pressure pain threshold
Diagnostic Test: Patient Health Questionnaire 9 — The Patient Health Questionnaire 9 (PHQ-9), a validated and internationally used health questionnaire, will also be completed twice at the first study day before the sex hormone therapy is initiated and during the last study day in month 6. The questionnaire consists of 9 items on the topic of mental well-being.
Diagnostic Test: Hormone concentrations — Blood concentrations of the following laboratory parameters will be determined:
  * Follicle stimulating hormone (FSH)
  * Luteotropic hormone (LH)
  * Prolactin (PRL)
  * Oestradiol (E2)
  * Sex hormone-binding globulin (SHBG)
  * Testosterone

SUMMARY:
It is known from the literature that women and men differ in their perception of pain. Why this is the case has not been conclusively clarified. Sex hormones could have a significant influence on this. The study team suspects that the classic hormone status of women is responsible for the lower pain threshold compared to men.

People undergoing gender affirming therapy receive biologically opposite-sex hormones in order to adapt their external appearance as well as their voice, emotional life etc. to the desired gender. The aim of this study is to longitudinally record whether the intake of opposite-sex sex hormones leads to a change in pain and perception thresholds in this patient collective. To this end, potential study participants will be informed about the study and asked whether they would like to participate before the start of hormone therapy during their first visit to the transgender outpatient clinic.

If consent is given, a questionnaire on mental health (PHQ 9), a blood sample to determine the hormone status and the first QST (quantitative sensory testing) measurement are then carried out. The second measurement with blood sampling takes place 3-4 weeks after the first measurement. The 3rd and 4th measurements with blood sampling are taken 3 and 6 months respectively after the first measurement. The PHQ 9 is measured again at the time of the last measurement. Study participation ends after a total of 6 months. The blood samples, the PHQ 9 and the QST measurements have no influence on the treatment of the study participants.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Assigned female at birth (AFAB)
* Diagnosed gender identity disorder/gender dysphoria and planned therapy with testosterone OR
* ≥ 18 years of age
* Assigned male at birth (AMAB)
* Diagnosed gender identity disorder/ gender dysphoria and planned therapy with estradiol

Exclusion Criteria:

* Any sex hormone intake during the last 6 months
* Acute or chronic pain
* Polyneuropathy
* Diagnosis of alcohol or drug addiction
* BMI under 18 or over 35
* Pregnancy
* Breastfeeding
* Pharmacological analgesic therapy within the previous 7 days before each examination
* History of significant trauma or surgery to the hands with residual neurological deficit or pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult participants, who must meet all of the prespecified inclusion criteria to be eligible for inclusion in the study and must not meet any of the prespecified exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Cold detection threshold | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  °C (Arithmetic mean after 3 measurement repetitions) With the Limits Method, the perception and pain thresholds are recorded as the first detected stimulus in the context of increasing stimulus intensities. This test will be performed with the Thermal Sensory Analyzer (TSA II, Medoc).
  A thermode equipped with a Peletier element and a cooling water supply is placed on the skin. Then the following parameters are determined using the Limits method:
  * Cold detection thresholds
  * Heat detection thresholds
  * Thermal difference thresholds for the detection of paradoxical heat sensations The contact area of the respective thermodes is 9.0 cm². By pressing a stop switch, which is connected to a computer unit, a threshold value determination can be made after a continuous ascending or descending temperature range with the thermode contact area, starting from a base temperature of 32°C. The temperature changes at a rate of 1°C/s.
Warm detection threshold | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  °C (Arithmetic mean after 3 measurement repetitions)
  With the Limits Method, the perception and pain thresholds are recorded as the first detected stimulus in the context of increasing stimulus intensities. This test will be performed with the Thermal Sensory Analyzer (TSA II, Medoc).
  A thermode equipped with a Peletier element and a cooling water supply is placed on the skin. Then the following parameters are determined using the Limits method:
  * Cold detection thresholds
  * Heat detection thresholds
  * Thermal difference thresholds for the detection of paradoxical heat sensations The contact area of the respective thermodes is 9.0 cm². By pressing a stop switch, which is connected to a computer unit, a threshold value determination can be made after a continuous ascending or descending temperature range with the thermode contact area, starting from a base temperature of 32°C. The temperature changes at a rate of 1°C/s.
Thermal sensory limen | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  °C With the Limits Method, the perception and pain thresholds are recorded as the first detected stimulus in the context of increasing stimulus intensities. This test will be performed with the Thermal Sensory Analyzer (TSA II, Medoc).
  A thermode equipped with a Peletier element and a cooling water supply is placed on the skin. Then the following parameters are determined using the Limits method:
  * Cold detection thresholds
  * Heat detection thresholds
  * Thermal difference thresholds for the detection of paradoxical heat sensations The contact area of the respective thermodes is 9.0 cm². By pressing a stop switch, which is connected to a computer unit, a threshold value determination can be made after a continuous ascending or descending temperature range with the thermode contact area, starting from a base temperature of 32°C. The temperature changes at a rate of 1°C/s.
Paradoxical heat sensation | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Number of Paradoxical heat sensation out of 3
  The paradoxical heat sensations (PHS) can occur during the determination of the TSL (thermal sensory limen) by thrice alternating cold and warm stimuli. A paradoxical heat sensation occurs when the patient expresses heat perceptions during an actual cold stimulus, contrary to what is indicated by the software, or vice versa. In the aforementioned thermal threshold measurement, alternating high and low temperatures are set on the thermode. The study participant does not know the sequence and must recognize the respective tendency. Alternating the temperature changes is done without resetting the initial temperature. PHS has no unit, it is given as a number: PHS 0; 1; 2 or 3, depending on the number of false temperature perceptions.
Cold pain threshold | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  °C (Arithmetic mean after 3 measurement repetitions) With the Limits Method, the perception and pain thresholds are recorded as the first detected stimulus in the context of increasing stimulus intensities. This test will be performed with the Thermal Sensory Analyzer (TSA II, Medoc).
  A thermode equipped with a Peletier element and a cooling water supply is placed on the skin. Then the following parameters are determined using the Limits method:
  * Cold detection thresholds
  * Heat detection thresholds
  * Thermal difference thresholds for the detection of paradoxical heat sensations The contact area of the respective thermodes is 9.0 cm². By pressing a stop switch, which is connected to a computer unit, a threshold value determination can be made after a continuous ascending or descending temperature range with the thermode contact area, starting from a base temperature of 32°C. The temperature changes at a rate of 1°C/s.
Heat pain threshold | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  °C (Arithmetic mean after 3 measurement repetitions) With the Limits Method, the perception and pain thresholds are recorded as the first detected stimulus in the context of increasing stimulus intensities. This test will be performed with the Thermal Sensory Analyzer (TSA II, Medoc).
  A thermode equipped with a Peletier element and a cooling water supply is placed on the skin. Then the following parameters are determined using the Limits method:
  * Cold detection thresholds
  * Heat detection thresholds
  * Thermal difference thresholds for the detection of paradoxical heat sensations The contact area of the respective thermodes is 9.0 cm². By pressing a stop switch, which is connected to a computer unit, a threshold value determination can be made after a continuous ascending or descending temperature range with the thermode contact area, starting from a base temperature of 32°C. The temperature changes at a rate of 1°C/s.
Mechanical detection threshold | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  mN (geometric mean of 5 even suprathreshold and 5 even subthreshold stimulus strengths)
  The mechanical detection threshold is measured with a set of standardized von Frey filaments. The von Frey filaments used in this test are glass fiber filaments with different diameters and varying lengths and with a spherical contact surface of approximately 0.5 mm diameter. The set used for the test consists of filaments with the strengths 0.25, 0.5, 1, 2, 4, 8, 16, 32, 64, 128, 256 and 512 mN. The contact time on the skin surface should be about 2 s during testing. To determine the tactile detection threshold, the geometric mean of 5 straight suprathreshold and subthreshold stimulus strengths is determined using a modified Levels method.
Mechanical pain threshold | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  mN (geometric mean of 5 even suprathreshold and 5 even subthreshold stimulus strengths) Needle stimulators (Pinprick) are used to determine the mechanical pain threshold. The models used consist of blunt needles with a fixed stimulation intensity of 8, 16, 32, 64, 128, 256 and 512 mN and a blunt circular skin contact surface with a diameter of 0.25 mm. The individual needle stimulators (pinpricks) are applied in 5 series of ascending and descending stimulus intensity with a skin contact time of about 1-2 s at a perpendicular angle to the skin. Likewise in this test, the actual mechanical pain threshold is calculated according to the Levels method as the geometric mean of 5 just above-threshold and 5 just below-threshold stimulus intensities.
Mechanical pain sensitivity | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Geometric mean of all numeric values (scale 1-100) Needle stimulators (Pinprick) are used to determine the mechanical pain threshold. The models used consist of blunt needles with a fixed stimulation intensity of 8, 16, 32, 64, 128, 256 and 512 mN and a blunt circular skin contact surface with a diameter of 0.25 mm. The individual needle stimulators (pinpricks) are applied in 5 series of ascending and descending stimulus intensity with a skin contact time of about 1-2 s at a perpendicular angle to the skin. Likewise in this test, the actual mechanical pain threshold is calculated according to the Levels method as the geometric mean of 5 just above-threshold and 5 just below-threshold stimulus intensities.
Dynamic mechanical allodynia | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Geometric mean of all numeric values (scale 1-100) A set consisting of the previously described needle stimulators, a cotton swab, a soft brush and a cotton ball will be used to determine the mechanical pain sensitivity of the skin and to detect the presence of any dynamic mechanical allodynia to light touch stimuli. Stimulus-response behaviours to needle stimuli and primarily non-painful, light touch stimuli are sequenced and evaluated. Subjects are asked to rate the perception of the stimulus on a numerical rating scale from 0 to 100 (0= no pain; 100= most pain imaginable). In the same test procedure, the extent of any dynamic mechanical allodynia is also determined, using the cotton ball (3 mN), cotton swab (100 mN) and standardised brush (Somedic, Sweden; 200-400 mN). These 3 tactile stimuli are stroked over the subject's skin by the examiner for about 2 s for at least 2 cm. Again, the subjects rate the stimulus on a numerical scale from 0 to 100.
Wind-up ratio | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Wind-up quotient (Sensation intensity of the stimulus series 1Hz/single stimulus) Needle stimulators with an intensity of 256 mN are used to determine the wind-up phenomenon. To determine wind-up, the sensitivity of the skin to a single stimulus is compared with that to a series of stimuli (10 needle stimuli) in the test area. The subject rates on a numerical pain scale the applied stimuli, i.e., the single stimulus and the entire stimulus series. The application of the single stimulus followed by the stimulus series is repeated 5 times. The wind-up quotient is calculated from the ratio of the perceived pain intensity over the stimulus series divided by the pain intensity after the single stimuli.
Vibration detection threshold | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Arithmetic mean after 3 measurement repetitions on a 8/8 scale Rydel-Seiffer tuning fork A Rydel-Seiffer tuning fork with a vibration frequency of 64 Hz and an 8/8 scale is used to determine the vibration threshold. To check the threshold values the struck and vibrating tuning fork is placed on the test area, preferably over a bony contact point such as the ankle. The test person indicates when he or she no longer feels the vibrations of the tuning fork. For this point in time, the stimulus intensity is recorded on the scale of the tuning fork. After determining the vibration threshold 3 times, the arithmetic mean of the threshold values can be calculated.
Pressure pain threshold | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  kPa (Arithmetic mean after 3 measurement repetitions) The measurement of the pressure pain threshold is carried out with the aid of a pressure algometer, on a blunt rubberized contact surface of about 1 cm², with which pressure of 0 to 2000 kPa can be applied. The pressure is gradually increased at a rate of 0.5 kg/cm²-s. The pressure pain threshold is documented as the value in Kpa at which the perception of pressure quality first changes to a painful sensory impression. The pressure pain threshold is calculated as an arithmetic mean after 3 repeated measurements.
Temperature of the skin | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  °C
  The temperature of the skin will be measured with a temperature probe.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 | At the time of enrollment and on the last study day after 6 months.
  Consists of 9 items concerning patient mental well-being. The EQ-5D-5L, a validated and internationally used health questionnaire, will also be completed twice at the first study day before the sex hormone therapy is initiated and during the last study day in month 6. It consists of a page with questions on mobility, self-care, usual activities, pain/discomfort and anxiety/depression as well as an assessment of one's own state of health on a scale of 1-100 (100 = best health you can imagine).
Hormone concentrations (follicle stimulating hormone) | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Laboratory measurement of follicle stimulating hormone (FSH) in mIU/mL
Hormone concentrations (luteotropic hormone) | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Laboratory measurement of luteotropic hormone (LH) in mIU/mL
Hormone concentrations (prolactin) | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Laboratory measurement of prolactin (PRL) in ng/mL
Hormone concentrations (oestradiol) | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Laboratory measurement of oestradiol (E2) in pg/mL
Hormone concentrations (sex hormone-binding globulin) | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Laboratory measurement of sex hormone-binding globulin (SHBG) in nmol/L
Hormone concentrations (testosterone) | At the time of enrollment and after 3-4 weeks, 3 months and 6 months.
  Laboratory measurement of testosterone in ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kimberger, Prof., Principal Investigator — Medical University of Vienna, Dept. of Anaesthesiology, Critical Care and Pain Medicine
Locations (1):
- Mecial University of Vienna, Vienna, Vienna, Austria